CLINICAL TRIAL: NCT04605835
Title: Ultrasonic Visualization of Renal Function Damage and Urodynamic Disorders for Obstructive Uropathies in Children
Brief Title: Ultrasonic Visualization of Obstructive Uropathies in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samarkand State Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DGU 20200967
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Uropathy
Keywords: obstructive uropathy; children; ultrasound; Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: 484 children with congenital obstructive uropathies
  Interventions: Diagnostic Test: ULTRASONIC VISUALIZATION OF OBSTRUCTIVE UROPATHIES IN CHILDREN.

INTERVENTIONS:
Diagnostic Test: ULTRASONIC VISUALIZATION OF OBSTRUCTIVE UROPATHIES IN CHILDREN. — The purpose of this study was to develop proposals and recommendations for improving the safety of urological examination of children with obstructive uropathy by using Doppler ultrasound. Based on the results of a comprehensive urological examination of 665 children with congenital ureteral obstruction, a program for scoring the results of ultrasound examination has been developed, which allows using the safest and most informative methods to reliably determine the functional state of the renal parenchyma and the degree of urodynamic disorders in children with obstructive uropathy.

SUMMARY:
The purpose of this study was to develop proposals and recommendations for improving the safety of urological examination of children with obstructive uropathy by using Doppler ultrasound. Based on the results of a comprehensive urological examination of 665 children with congenital ureteral obstruction, a program for scoring the results of ultrasound examination has been developed, which allows using the safest and most informative methods to reliably determine the functional state of the renal parenchyma and the degree of urodynamic disorders in children with obstructive uropathy.

DETAILED DESCRIPTION:
Relevance. The prevalence of congenital diseases of the genitourinary system is 0.5-7.5 per 1000 newborns; The high prevalence reflects the medical and social significance of the problem and determines the need to search for highly informative and safe diagnostic methods for the child's body, providing timely treatment, restoration of the somatic and social status of children.

Purpose. Development of proposals and recommendations to improve the safety of urological examination of children with obstructive uropathy.

Material and methods. The study is based on the analysis of the results of diagnosis and treatment of 655 children with congenital obstruction of the upper urinary tract. The complex of urological examination included clinical, laboratory, morphological, radiological, ultrasound research methods.

ELIGIBILITY:
Inclusion Criteria:

* 655 children with congenital obstruction of the upper urinary tract

Exclusion Criteria:

* none

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 60 in children with obstructive uropathies (30 children with congenital hydronephrosis and 30 children with congenital ureterohydronephrosis).
Sampling Method: Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasonic visualization of renal function damage and urodynamic disorders for obstructive uropathies in children. | up to 36 months
  The purpose of this study was to develop proposals and recommendations for improving the safety of urological examination of children with obstructive uropathy by using Doppler ultrasound. Based on the results of a comprehensive urological examination of 665 children with congenital ureteral obstruction, a program for scoring the results of ultrasound examination has been developed, which allows using the safest and most informative methods to reliably determine the functional state of the renal parenchyma and the degree of urodynamic disorders in children with obstructive uropathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Samarkand State Medical Institute, Samarkand, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: American Journal of Roentgenology — https://www.arrs.org/ARRSLIVE/Publications